CLINICAL TRIAL: NCT04515706
Title: Safety, Tolerability, Efficacy of Iguratimod in Systemic Sclerosis
Brief Title: Iguratimod in Systemic Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IGU
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Systemic Sclerosis, Diffuse
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — iguratimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iguratimod (Experimental): Iguratimod 25 twice a day (bid) on Week 1-48.
  Interventions: Drug: Iguratimod
- Placebo (Placebo Comparator): Placebo twice a day (bid) on Week 1-24, and Iguratimod 25 twice a day (bid) on Week 25-48.
  Interventions: Drug: Iguratimod; Drug: Placebo

INTERVENTIONS:
Drug: Iguratimod — Iguratimod is an anti-rheumatic drug that approved for treating rheumatoid arthritis in East Asia. Recent data reveal its independent anti-fibrosis effect.
Drug: Placebo — Placebo of Iguratimod
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of iguratimod in adult subjects with diffuse cutaneous systemic sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic sclerosis (SSc), as classified using the 2013 American College of Rheumatology/ European Union League Against Rheumatism classification of SSc.
* Diffuse Cutaneous Systemic Sclerosis (dcSSc) as defined by 2001 LeRoy and Medsger Disease duration ≤ 3 years (defined as time from the first non-Raynaud phenomenon manifestation).
* Agree to use effective contraception during the study period (women of childbearing age).
* Smokers agreed to quit smoking during the study.
* Ability to provide informed consent.

Exclusion Criteria:

* The following drugs have been used within one month before screening: including TNF-α inhibitors (continuous use for more than 14 days), IL-6 inhibitors, abatacept (continuous use for more than 14 days), JAK inhibitors (continuous use for more than 14 days).
* Used rituximab within 3 months before screening.
* SSc with tumor.
* People with various lung infections, asthma or other lung diseases such as bronchiectasis.
* For patients with severe heart, liver, kidney and other important organ dysfunction, the evaluation criteria are as follows: ALT or AST is greater than 2 times the upper limit of normal, or total bilirubin rises twice; CPK>400; Renal crisis, or hypertension of various causes (≥160/100mmHg) is not controlled; Creatinine clearance rate <30ml/min; White blood cell count<3×109/L; Hemoglobin <80g/L; Platelet count<60×109/L; Heart function level III-IV; PaO2<50mmHg in resting state; FEV1/FVC<0.7.
* In the period of acute or chronic infection (not including finger ulcer combined infection).
* A history of peptic ulcer or bleeding within 6 months before screening.
* People with allergies or multiple drug allergies.
* People with mental illness or other reasons who cannot cooperate with treatment.

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience Grade 3 or Higher Adverse Events That Occur at or Before Week 24 | Week 24
  Primary outcome is met if any participants experience a grade 3 or higher event prior to Week 24. A grade 3 AE would constitute as "severe". Grading was following using CTCAE v 4.03.

SECONDARY OUTCOMES:
Number of Grade 3 (Severe) or Higher Adverse Events That Occur Throughout the Study | Week 12, 24, 36, and 48
  Grade 3 or higher adverse events (AEs) assessed throughout the study ( 48 weeks). A grade 3 AE would constitute as "severe". Grading was following using CTCAE v 4.03.
Number of Grade 2 (Moderate) or Higher Adverse Events That Occur Throughout the Study | Week 12, 24, 36, and 48
  Grade 2 or higher assessed 12 weeks apart. Grade 2 AEs are determined as " moderate". Grading was performed following CTCAE v 4.03 guidance.
Provisional American College of Rheumatology Combined Response Index (CRISS) Systemic Sclerosis | Week 12, 24, and 48
  CRISS components included the following domains: modified Rodnan skin score, forced vital capacity percent predicted, Physician Global Assessment, Patient Global Assessment, and Health Assessment Questionnaire Disability-Index. An algorithm determines the predicted probability of improvement from baseline by incorporating change in the mRSS, FVC percent predicted, Physician and Patient Global Assessments, and HAQ-DI. The outcome is a continuous variable between 0.0 and 1.0 (0 - 100%). A cut-off at 0.6 in the predicted probability of being improved has yielded the smallest misclassification error. Subjects are not considered improved if, between Visit 1 and 6, they develop new: 1) renal crisis; 2) decline in FVC% predicted by 15% (relative) from baseline and confirmed after 1 month; or 3) left ventricular failure (systolic ejection fraction < 45%) or pulmonary artery hypertension. Higher CRISS scores indicates improvement.
Scleroderma Clinical Trials Consortium Damage Index | Week 24, 48
  A damage Index (DI) in systemic sclerosis, including musculoskeletal and skin, vascular, gastrointestinal, respiratory and cardiovascular damage caused by SSc.
Change in Modified Rodnan Skin Score (mRSS) | Week 12, 24, 36, and 48
  The Modified Rodnan Skin Score (mRSS) is a measure of skin thickness. Skin thickness in 17 anatomic areas was rated on a 0-3 scale and scores are summed to obtain the mRSS (range from 0 - 51), with higher mRSS scores indicating worse disease activity
Change in Skin Thickness | Week 24, 48
  The skin thickness of fingers and palms would be measured by high frequency echo. detector.

IPD SHARING:
Plan to Share IPD: No